CLINICAL TRIAL: NCT05193591
Title: Evaluation of Anti-C1s, Anti-HMGB1 and Anti-C1q Autoantibodies in the Pathogenesis for Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Anti-C1s, Anti-HMGB1 and Anti-C1q Autoantibodies in Systemic Lupus Erythematosus (DYSALARM-322)
Acronym: DYSALARM-322
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0388; 2021-A02672-39 (Other: ID RCB)
Record Dates: First submitted 2021-12-02; First posted 2022-01-18 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One serum sample per patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Autoantibodies evaluation in lupus — Biological analysis: anti-C1s, anti-HMGB1 and anti-C1q autoantibodies; C1s, HMGB1 and C1q proteins.
  Purification of patients' autoantibodies (anti-C1s, anti-HMGB1and anti-C1q). Identification of the molecular targets recognized by anti-C1s, anti-HMGB1 and anti-C1q autoantibodies purified from the SLE patients' serum.

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by the production of multiple autoantibodies and accumulation of immune complexes resulting in systemic inflammatory response and tissue damage.

Dysfunction of proteins initially known to initiate the classical pathway for complement activation (C1q and C1s), and their functional interference with the multifunctional protein HMGB1 (High-Mobility Group Box 1), appears to be associated with SLE. On the other hand, C1s, HMGB1 and C1q can be targeted by anti-C1s, anti-HMGB1 and anti-C1q autoantibodies from lupus patients, whose functional impact remains to be explored, in particular for non-canonical functions, independent of the complement activation cascade.

Studies are needed to investigate the pathogenic role of these autoantibodies in SLE, including possible interference with the inactivation of HMGB1.

This project plans to investigate the role of anti-C1s, anti-HMGB1 and anti-C1q autoantibodies in the pathogenesis of Systemic Lupus Erythematosus. This pilot study will be performed for 30 patients with active SLE on serum, realized for routine patient care. The investigators will identify the molecular targets recognized by anti-C1s, anti-HMGB1 and anti-C1q autoantibodies purified from the SLE patients' serum. The investigators will also explore the functional role of these purified autoantibodies.

DETAILED DESCRIPTION:
Regarding the exploration of anti-C1s autoantibodies purified from the SLE patients' serum, the investigators will evaluate their effects on the formation of the C1r2C1s2 tetramer and interaction with C1q and their effects on the esterase activity of C1s.

Regarding the exploration of anti-HMGB1 autoantibodies purified from the SLE patients' serum, the investigators will evaluate their effects on the binding of HMGB1 to its RAGE receptor and their effects on the binding of HMGB1 to C1q.

Regarding the exploration of anti-C1q autoantibodies purified from the SLE patients' serum, the investigators will evaluate their effects on the binding of C1q to its receptors and to the C1r2C1s2 tetramer and their effects on the activation of the classical Complement pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Weight ≥ 40 Kg
* Patients who have valid health insurance
* Patients with lupus diagnosis criteria (EULAR-ACR-2019)
* Active lupus nephritis defined by SLEDAI score >5 and joint and/or kidney involvement.

Exclusion Criteria:

* Patient protected by law (minors, pregnant or breastfeeding women, subject under guardianship or curatorship, deprived of liberty or enforced hospitalized, under administrative or judicial supervision).
* Patient on dialysis or on plasma exchange.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients: 30 patients with active lupus (joint and/or kidney involvement). SLE patients will be enrolled from departments of Internal Medicine (Grenoble University Hospital, France) and Nephrology (Conception University Hospital Marseille, France).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Quantification of anti-C1s autoantibodies purified from the serum of lupus patients with active disease, targeting N-terminal, C-terminal domains and C1s protease mutants. | Inclusion is the only visit (only one time point)
  Analysis: Levels of anti-C1s autoantibodies targeting N-terminal, C-terminal domains and C1s protease mutants by homemade ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal DUMESTRE-PERARD, Professor, Principal Investigator — Grenoble Alpes University Hospital
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - AP-HM_Hôpital de la Conception, Marseille

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunkelberger JR, Song WC. Complement and its role in innate and adaptive immune responses. Cell Res. 2010 Jan;20(1):34-50. doi: 10.1038/cr.2009.139. Epub 2009 Dec 15. PMID 20010915
- [Background] Macedo AC, Isaac L. Systemic Lupus Erythematosus and Deficiencies of Early Components of the Complement Classical Pathway. Front Immunol. 2016 Feb 24;7:55. doi: 10.3389/fimmu.2016.00055. eCollection 2016. PMID 26941740
- [Background] Schaper F, Westra J, Bijl M. Recent developments in the role of high-mobility group box 1 in systemic lupus erythematosus. Mol Med. 2014 Mar 13;20(1):72-9. doi: 10.2119/molmed.2014.00019. PMID 24531837
- [Background] Yeo JG, Leong J, Arkachaisri T, Cai Y, Teo BH, Tan JH, Das L, Lu J. Proteolytic inactivation of nuclear alarmin high-mobility group box 1 by complement protease C1s during apoptosis. Cell Death Discov. 2016 Sep 12;2:16069. doi: 10.1038/cddiscovery.2016.69. eCollection 2016. PMID 27648302
- [Background] He S, Lin YL. In vitro stimulation of C1s proteolytic activities by C1s-presenting autoantibodies from patients with systemic lupus erythematosus. J Immunol. 1998 May 1;160(9):4641-7. PMID 9574573
- [Background] Moroni G, Quaglini S, Radice A, Trezzi B, Raffiotta F, Messa P, Sinico RA. The value of a panel of autoantibodies for predicting the activity of lupus nephritis at time of renal biopsy. J Immunol Res. 2015;2015:106904. doi: 10.1155/2015/106904. Epub 2015 Feb 26. PMID 25815344
- [Background] Lintner KE, Wu YL, Yang Y, Spencer CH, Hauptmann G, Hebert LA, Atkinson JP, Yu CY. Early Components of the Complement Classical Activation Pathway in Human Systemic Autoimmune Diseases. Front Immunol. 2016 Feb 15;7:36. doi: 10.3389/fimmu.2016.00036. eCollection 2016. PMID 26913032